CLINICAL TRIAL: NCT04175418
Title: The Effects of a Supervised Exercise Program Versus Online Education Program to Increase Physical Activity in Patients With Multiple Sclerosis
Brief Title: The Effects of Two Different Types of Exercise Programs to Increase Physical Activity in Patients With MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Prof.Dr.Mazhar Osman Mental Health and Psychiatric Diseases Education, Research Hospital (Unknown)
Responsible Party: Principal Investigator, Gamze Öztürk, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IU-C
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Rehabilitation; Physical Activity; Exercise
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised Exercise Program Group (Experimental): Participants in the supervised exercise group were included to a program that consisted of 16 individual physiotherapist supervised sessions (two 60-minutes sessions/week), which were prepared to improve physical activity.
  Interventions: Other: Supervised Exercise Program
- Online Education Program Group (Experimental): Participants in the online education group were included to a program that consisted of 16 online sessions (two 60-minutes sessions/week), which were prepared to improve physical activity.
  Interventions: Other: Online Education Program

INTERVENTIONS:
Other: Supervised Exercise Program — The exercise program in this group includes aerobic (walking) training and exercises to strengthen the upper and lower extremities and trunk muscles.
  Arms: Supervised Exercise Program Group
Other: Online Education Program — The exercise program in this group includes aerobic (walking) training and home exercises to strengthen the upper and lower extremities and trunk muscles.
  Arms: Online Education Program Group

SUMMARY:
Multiple Sclerosis (MS) is a chronic, inflammatory, neurodegenerative, autoimmune disease of the central nervous system. It is thought that MS, which is one of the main causes of non-traumatic neurological dysfunction in young adults, affects approximately two and a half million people worldwide. The annual cost caused by MS is reported to be between $ 8,528 and $ 54,244 per patient. Due to the destruction of the central nervous system, MS has a wide range of sensory, motor, cerebellar and cognitive dysfunctions. These dysfunctions may lead to a limitation of physical activity in people with MS. In addition, people with MS may limit their physical activity because they fear the worsening of their symptoms. Physical inactivity and sedentary life style are thought to be among the reasons that increase the risk of developing chronic diseases such as cancer, hypercholesterolemia, hypertension, arthritis, osteoporosis, obesity, type 2 diabetes, depression and cardiovascular diseases in people with MS. It is reported that these chronic diseases secondary to MS increase mortality by 1.7 times. In addition, these diseases have been associated with increased disability, decreased quality of life, and hospitalization. Physical inactivity can increase disability and mortality by aggravating health problems caused by the disease. For this reason, it is emphasized that there should be studies to increase physical activity in people with MS. Studies have shown that physical activity improves muscle strength, aerobic capacity, gait and balance and reduces fatigue in people with MS. In addition, it is stated that physical activity increases self-efficacy and improves positive perspective in patients with MS. When the literature is examined, it is seen that there are studies about physical activity in MS but they have methodological limitations. There are a limited number of studies on the effectiveness of the programs planned to increase the level of physical activity. The aim of our study was to investigate the effects of physical activity program and online training program on physical activity in patients with MS.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Multiple Sclerosis
* Being between 25 and 60 age range
* Not having attacks during last 3 months
* Having ≤ 5.5 Expanded Disability Status Scale
* Not having received physiotherapy and rehabilitation sessions for at least 3 months
* Having internet access

Exclusion Criteria:

* Pregnancy
* Blurred vision
* Use of assistive devices for ambulation
* Having another diagnosis rather than Multiple Sclerosis

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
The Leisure-Time Exercise Questionnaire | 1-3 minutes
  It is a self-reported leisure-time exercise questionnaire which consists of 2 parts. The first part seeks information about the number of times one engages in mild, moderate and strenuous leisure-time exercise bouts of at least 15 min duration in a typical week. The weekly frequency of mild, moderate and strenuous exercise bouts are multiplied by 3, 5, and 9 metabolic equivalents (METs) and the total score is recorded. Second part seeks information about frequency of activity which is long enough to work up sweat in a typical week.
Pedometer | one week
  It is one of the objective methods used to evaluate physical activity. It is used to record the number of steps taken. The estimated step length is entered in the device and recorded as a step when the vertical swing of the body exceeds a certain threshold.

SECONDARY OUTCOMES:
6 Minute Walk Test | 6 minutes
  The 6-min walk test (6 MWT) is a submaximal exercise test that entails measurement of distance walked on a 30 meter course over a span of 6 minutes.
Multiple Sclerosis Walking Scale-12 | 3-5 minutes
  It is a scale consisting of 12 questions about mobility which is used to measure walking capacity. The limitations of walking in the last two weeks are questioned. Answers are scored between 1-5 (1 = almost none, 5 = excessive). A high score indicates that the ability to walk is affected or that the patient has difficulty in walking.
Fatigue Severity Scale | 3-5 minutes
  It is a scale that evaluates the fatigue of MS patients in daily functions. The assessment consists of 9 questions, each question is scored between 1 (strongly disagree) to 7 (strongly agree). The result score is the average value of nine questions. High score indicates increased fatigue severity
Multiple Sclerosis International Quality of Life Questionnaire | 5-7 minutes
  The scale consists of 31 questions in 6 sub-groups including physical status, symptoms, psychological status, self-esteem, relationship with friends, family and medical staff. The answers are scored between 0 and 5 and a score between 0 and100 is obtained. The higher the score, the higher the level of quality of life.
Brief International Cognitive Assessment for MS | 15 minutes
  The Brief International Cognitive Assessment for MS is composed of 3 parts.In these parts, data processing speed, verbal memory, and visual memory are evaluated.
Bioelectrical Impedance Analysis | 1-2 minutes
  It is a method that is based on measurement of body resistance with the aid of alternative electric current. Body components are calculated by this method.
Muscle Strength Test | 45 minutes
  The isokinetic dynamometer and handheld dynamometer are used to assess muscle strength. In this study, the isokinetic dynamometer will be used to evaluate the knee extensor and flexor concentric muscle strength and the handheld dynamometer will be used to evaluate upper extremity muscle strength including arm flexors, abductors, elbow flexors and lower extremity muscle strength including hip flexors and abductors.

CONTACTS AND LOCATIONS:
Overall Officials: Yonca Zenginler Yazgan, Ph.D, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)